CLINICAL TRIAL: NCT04836663
Title: A Open-label, Multicenter Phase II Study of TQ-B3525 Tablets in Subjects With PIK3CA and/or PIK3R1/2 Gene-altered Recurrent/Metastatic Advanced Gynecologic Tumors
Brief Title: A Study of TQ-B3525 Tablets in Subjects With PIK3CA and/or PIK3R1/2 Gene-altered Recurrent/Metastatic Advanced Gynecologic Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3525-II-03
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-04

CONDITIONS: Advanced Endometrial Cancer, Cervical Cancer and Ovarian Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Ovarian Neoplasms | interventions — TQ-B3525

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ-B3525 tablet (Experimental)
  Interventions: Drug: TQ-B3525 tablet

INTERVENTIONS:
Drug: TQ-B3525 tablet — TQ-B3525 tablet administered orally once a day. Each cycle is 28 days.

SUMMARY:
This is a study to evaluate the efficacy and safety of TQ-B3525 in subjects with recurrent / metastatic advanced endometrial cancer, cervical cancer and ovarian cancer with PIK3CA and / or PIK3R1 / 2 gene-altered (mutation or amplification). Endometrial cancer, cervical cancer and ovarian cancer are divided into three cohorts, each cohort administrated TQ-B3525 tablet orally once a day.

ELIGIBILITY:
Inclusion Criteria:

* 1. Pathologically confirmed malignant gynecological neoplasm. 2. Has PIK3CA and/or PIK3R1/2 Gene-altered. 3.Unresectable, locally advanced recurrent and/or metastatic tumors, has at least 1 measurable lesion.

  4.Failed with standard treatment or has no effective treatment. 5. 18 years and older, Eastern Cooperative Oncology Group(ECOG) performance status score of 0 to 1, Life expectancy ≥ 3 months.

  6. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the first administration.

  7.Understood and signed an informed consent form.

Exclusion Criteria:

* 1.Has untreated or active central nervous system metastases. 2.Has diagnosed and/or treated additional malignancy within 3 years prior to the first administration.

  3. Insufficient hematopoietic function of bone marrow. 4. Dysfunction of liver and kidney. 5. Bleeding risk. 6. Dysfunction of gastrointestinal tract. 7.Dysfunction of heart and cerebral vessels. 8.Has received PI3K, AKT, mTOR inhibitor. 9.Has participated in other clinical trails within 30 days. 10. Has received surgery, or unhealed wounds within 4 weeks before the first administration.

  11. Has received organ grafting, or hematopoietic stem cell transplantation within 60 days before the first administration, or host versus graft reaction.

  12. The patients required immunosuppressor, or the whole-body, or absorbable local hormone therapy for immunosuppression purposes and continued to use within 7 days before the initial administration (daily dose of glucocorticoid <10 mg, except metacortandracin or other therapeutic hormones and so on).

  13. Has active infections. 14. Has human immunodeficiency virus (HIV). 15. Pregnant or lactating women. 16. Has psychotropic substances abuse or a mental disorder. 17. Has other conditions that make it inappropriate for the patient to be enrolled based on investigator's opinion.

  18. Patient's compliance is inadequate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) assessed by Independent Review Committee | up to 48 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR) based on IRC.

SECONDARY OUTCOMES:
Overall response rate (ORR) assessed by Investigator | up to 48 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR) assessed by investigator.
Disease control rate（DCR） | up to 48 weeks
  Percentage of subjects achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of disease remission (DOR) | up to 48 weeks
  The time from the first evaluation of the subject as CR or PR to the first evaluation of the subject as PD or death (whichever occurs first).
Progression-free survival (PFS) | up to 48 weeks
  PFS was defined as the time from the date of study enrollment to the date of the first of the following events, objective disease progression or death due to any cause.
Overall survival (OS) | up to 72 weeks
  OS defined as the time from the first dose to death from any cause. Survival time was censored at the date of last contact for patients who were still alive or lost to follow-up.
DOR rate (≥ 6 months) (percentage of subjects with disease remission duration ≥ 6 months) | up to 48 weeks
  The percentage of subjects achieving CR or PR was recorded for the first time to 6 months after the first time of objective tumor progression or death due to any cause (whichever occurred first) was recorded.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital Medical School Zhejiang University, Hangzhou, Zhejiang